CLINICAL TRIAL: NCT00587873
Title: Sequential Administration of Oral 6-Thioguanine (6-TG) After Methotrexate (MTX) in Patients With Relapsed Hodgkin's Disease (Phase II)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Tanya Trippett, MD, Memorial Sloan-Kettering cance Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 94-030
Record Dates: First submitted 2007-12-26; First posted 2008-01-08 (Estimated); Last update posted 2009-06-12 (Estimated); Status verified 2009-06

CONDITIONS: Hodgkin's Disease
Keywords: Relapsed; Hodgkin's Disease; Methotrexate; 6-Thioguanine; 94-030
MeSH Terms: conditions — Hodgkin Disease; Recurrence | interventions — Methotrexate; Leucovorin; Thioguanine

ARMS (1):
- 1 (Experimental): MTX, 6-TG, and Leucovorin combination
  Interventions: Drug: Methotrexate; Drug: Leucovorin calcium; Drug: 6-Thioguanine

INTERVENTIONS:
Drug: Methotrexate — MTX 6mg/m2 given IV bolus, followed by 24mg/m2 given in 24hrs continuous infusion
  Other Names: MTX
Drug: Leucovorin calcium — 5 mg orally at 12 hours after the end of MTX infusion then every 12 hrs for a total of 3 doses.
Drug: 6-Thioguanine — 6-TG 300 mg/m2 PO as a single oral dose
  Other Names: 6-TG

SUMMARY:
The objective of this study is to determine the incidence of complete and partial response and the duration of response in patients with recurrent or resistant Hodgkin's disease (HD) treated with sequential administration of oral 6-Thioguanin (6-TG) after IV Methotrexate (MTX).

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologic proof of HD who are in relapse and have failed > or = to 2 prior chemotherapy regimens.
* Patients must have a life expectancy of at least 8 weeks.
* All patients must have ECOG performance level rating of < or = to 2.
* Patients or their parents (guardian) must sign an informed consent indicating that they are aware of the investigational nature of the study.
* Patients must have recovered from the toxic effects of prior therapy before entering this study or at least 2 weeks should have elapsed since the end of last course of CT.
* Patients must have adequate liver function (bilirubin < or = to 2.0 mg/dl, SGOT less than 1.5 times normal (unless it is due to disease), adequate renal function (creatinine < or = to 1.5 mg/dl, creatinine clearance > or = to 60 ml/min/1.73 m2).
* Patients should have a granulocyte count > or = to 500/gL and a platelet count > or = to 100,000/uL (unless due to disease involvement of the bone marrow).
* Male and female patients of child-bearing age should use effective methods of contraception, if sexually active.

Exclusion Criteria:

* Patients with active infections or significant medical conditions other than their malignancy shall be excluded.
* Patients with HD who had prior MTX or 6-TG should be excluded.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 1994-03; Primary Completion 2003-12 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
To determine the incidence of complete and partial response and the duration of response in patients with recurrent or resistant Hodgkin's Disease (HD) treated with sequential administration of oral 6-Thioguanine (6-TG) after IV Methotrexate (MTX). | Conclusion of the study

SECONDARY OUTCOMES:
Define Toxicity of this sequential drug combination. | Conclusion of study

CONTACTS AND LOCATIONS:
Overall Officials: Tanya Trippett, MD, Principal Investigator — Memorial Sloan-Kettering Cancer Center/94-030
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Related Info — http://www.mskcc.org